CLINICAL TRIAL: NCT04455256
Title: Endoplasmic Reticulum Stress in Recurrent Pregnancy Loss
Brief Title: Evaluation of Endoplasmic Reticulum Stress in Patients With Recurrent Pregnancy Loss
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: tgk-xbp
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Pregnancy Loss; Endoplasmic Reticulum Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recurrent pregnancy loss group: Women between the ages of 18 and 45 who had a history of miscarriage under 3 weeks and above 22 weeks were included in this group.
  Interventions: Other: x box binding protein
- women who had healthy birth: Women between the ages of 18-45 who have not had a history of pregnancy loss and who have had at least one healthy birth and no known chronic diseases are included in this group.
  Interventions: Other: x box binding protein

INTERVENTIONS:
Other: x box binding protein — Serum value (pg / mL) of x box binding protein (XBP-1), which is one of the unfolded proteins indicating endoplasmic reticulum stress, is measured.

SUMMARY:
To evaluate endoplasmic reticulum stress in women with recurrent pregnancy loss and those who had healthy births in the same age group. The level of the unfolded protein X box binding protein 1 (XBP-1) is measured. It is aimed to show the effect of endoplasmic reticulum stress on recurrent pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* with three or more miscarriages before 20 th week of gestation
* had no chronic or acute inflammatory disease
* used no steroids, anti-inflammatory, or antioxidant medications

Exclusion Criteria:

* had inflammatory diseases
* had systemic disease
* Anatomical abnormalities, infectious, endocrine, or genetic etiologies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Loss of 3 or more pregnancy between the ages of 18 and 45 and women who have given at least 1 healthy birth in the same age group.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Show the effect of endoplasmic reticulum stress on recurrent pregnancy loss | 3 months
  Serum value (pg / mL) of x box binding protein (XBP-1), which is one of the unfolded proteins indicating endoplasmic reticulum stress, is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes